CLINICAL TRIAL: NCT02523001
Title: Urinary AQP2 Excretion in Hypercholesterolemic Patients as a Measure of Effect of Statin Therapy
Brief Title: Effect of Statin Treatment on Urinary AQP2 (uAQP2/01)
Acronym: uAQP2/01
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, piero portincasa, Professor of Medicine, PhD, University of Bari
Other Study IDs: uAQP2/01; MRAR08P011 (Other: Italian Agency of Drug (AIFA))
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Hypercholesterolemia; Diabetes Insipidus
MeSH Terms: conditions — Hypercholesterolemia; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood analyses (serum lipids, creatininemia, glucose, bilirubin) Urines (creatininuria, urinary AQP2)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Naïve-S: Patients with hypercholesterolemia starting statin treatment for primary or secondary prevention of cardiovascular diseases.
- ONC-S: Patients with hypercholesterolemia who had been treated with statin for at least one year and continued their previous therapy during the study period
- Naïve-MC: Patients with mild hypercholesterolemia either refusing initial statin treatment or intolerant to standard statin treatment and starting with monacolin K
- Naïve-Diet: Patients refusing an initial pharmacologic treatments and choosing the hypolipidic diet

SUMMARY:
The purpose of this study is to test the hypothesis that the function and/or regulation of urinary aquaporin 2 in hypercholesterolemic humans is affected by standard statin therapy, as compared with diet alone

DETAILED DESCRIPTION:
Statins are the first-line recommended pharmacological therapy in patients with dyslipidemias and play a key role in both primary and secondary prevention of coronary heart disease. By decreasing plasma total and low-density lipoprotein cholesterol (LDL-C) concentrations, statins decrease the risks for atherosclerotic cardiovascular disease and associated morbidity and mortality. Statins occupy part of the active binding site of 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) and inhibit its enzymatic activity in the liver, a key step leading to the reduction of cellular sterol pool. Statins also have beneficial effects on the vascular wall by stabilizing the atherosclerotic plaques, ameliorating impaired endothelial function, and reducing vascular inflammation.

Besides the well-known metabolic and cardiovascular effects, it has been recently shown that statins increase the plasma membrane expression of the renal water channels Aquaporin 2 (AQP2). Water reabsorption in the kidney connecting tubule and collecting duct is regulated by the antidiuretic hormone arginine vasopressin (AVP), which promotes plasma membrane expression of the water channe aquaporin 2 (AQP2), the rate-limiting step controlling reabsorption of water, thus urine concentration, in this segment of the nephron. The investigators reported a number of evidences showing that statins accumulate AQP2 at the apical membrane of collecting duct cells by a AVP-independent mechanism. The effect of statins on AQP2 is independent of classical cholesterol homeostasis but rather depends on depletion of mevalonate-derived intermediates of cholesterol synthetic pathways, i.e. isoprenoid intermediates, including farnesylpyrophosphate (FPP) and geranylgeranylpyrophosphate (GGPP).

Water balance disorders are often associated with defects of AQP2 trafficking. Nephrogenic Diabetes Insipidus (NDI) is characterized by the inability of the kidney to respond to AVP stimulation and is caused by either mutations in AQP2 or vasopressin type-2 receptor (AVPR2) genes. Mutations in the AVPR2 gene lead to X-linked NDI (X-NDI). This cause of 90% of all diagnosed congenital NDI cases.

Conventional treatment of X-NDI patients consists in low-sodium, low-protein diet and the administration on thiazide diuretics sometimes in combination with indomethacin or amiloride. Although these drugs cause some relief of X-NDI symptoms, they most often do not eliminate them. Due to the partial beneficial effect of conventional treatments, much effort has been spent in the past years to uncover new and alternative methods to induce antidiuresis in X-NDI patients.

In this regard, the investigators recently reported that statins, in particular fluvastatin, accumulate AQP2 at the apical membrane of collecting duct cells by a AVP-independent mechanism and increase water reabsorption in both wild type and X-NDI mice.

The effect of statins on AQP2 trafficking in humans, however, deserves further investigation, also considering the potential efficacy of statins in patients with X-NDI. This was the reason to embark on the present study in which the investigators monitored the time-dependent effects of statin therapy on the urine excretion of AQP2, diuresis and urine osmolality in a cohort of hypercholesterolemic subjects initiating simvastatin therapy for three months. Two other groups of patients serve as controls: patients already on statin treatment and patients choosing to undergo an initial program with a standard hypolipidemic "mediterranean" style diet.

ELIGIBILITY:
Inclusion criteria:

* patients on primary prevention requiring moderate reduction of LDL-cholesterol according to the ACC/AHA Guidelines
* age 40 to 75 years
* estimated 10-year ASCVD risk ≥7.5%

Exclusion criteria:

* concomitant type 1 or type 2 diabetes
* blood hypertension
* concomitant use of diuretics or other drugs interfering with simvastatin

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Behavioral: diet Drug: statins, as required according to the ACC/AHA guidelines Diagnostic: anthropometric data, abdominal and carotid ultrasonography, serum (lipids, renal function) and urinary (AQP2, osmolality) dosages at enrollment and during a 3-months follow up (week 0, 1, 4, 12)
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
uAQP2 | 0, 1, 4, 12 weeks
  Urinary AQP2 excretion during therapy (statin or diet)

SECONDARY OUTCOMES:
Cholesterolemia | 0, 1, 4, 12 weeks
  Serum cholesterol during therapy (statin or diet)

CONTACTS AND LOCATIONS:
Overall Officials: Piero Portincasa, Principal Investigator — University of Bari Medical School
Locations (1):
- Department of Biomedical Sciences Human Oncology - Clinica Medica "A. Murri", Bari, Italy

REFERENCES:
- [Background] Greenwood J, Steinman L, Zamvil SS. Statin therapy and autoimmune disease: from protein prenylation to immunomodulation. Nat Rev Immunol. 2006 May;6(5):358-70. doi: 10.1038/nri1839. PMID 16639429
- [Background] Pisitkun T, Shen RF, Knepper MA. Identification and proteomic profiling of exosomes in human urine. Proc Natl Acad Sci U S A. 2004 Sep 7;101(36):13368-73. doi: 10.1073/pnas.0403453101. Epub 2004 Aug 23. PMID 15326289
- [Background] Valenti G, Laera A, Pace G, Aceto G, Lospalluti ML, Penza R, Selvaggi FP, Chiozza ML, Svelto M. Urinary aquaporin 2 and calciuria correlate with the severity of enuresis in children. J Am Soc Nephrol. 2000 Oct;11(10):1873-1881. doi: 10.1681/ASN.V11101873. PMID 11004218
- [Background] Kanno K, Sasaki S, Hirata Y, Ishikawa S, Fushimi K, Nakanishi S, Bichet DG, Marumo F. Urinary excretion of aquaporin-2 in patients with diabetes insipidus. N Engl J Med. 1995 Jun 8;332(23):1540-5. doi: 10.1056/NEJM199506083322303. PMID 7537863
- [Background] Valenti G, Laera A, Gouraud S, Pace G, Aceto G, Penza R, Selvaggi FP, Svelto M. Low-calcium diet in hypercalciuric enuretic children restores AQP2 excretion and improves clinical symptoms. Am J Physiol Renal Physiol. 2002 Nov;283(5):F895-903. doi: 10.1152/ajprenal.00354.2001. PMID 12372764
- [Background] Wade JB. Statins affect AQP2 traffic. Am J Physiol Renal Physiol. 2011 Aug;301(2):F308. doi: 10.1152/ajprenal.00248.2011. Epub 2011 May 11. No abstract available. PMID 21561996
- [Background] Li W, Zhang Y, Bouley R, Chen Y, Matsuzaki T, Nunes P, Hasler U, Brown D, Lu HA. Simvastatin enhances aquaporin-2 surface expression and urinary concentration in vasopressin-deficient Brattleboro rats through modulation of Rho GTPase. Am J Physiol Renal Physiol. 2011 Aug;301(2):F309-18. doi: 10.1152/ajprenal.00001.2011. Epub 2011 Apr 20. PMID 21511701
- [Background] Grunfeld JP, Rossier BC. Lithium nephrotoxicity revisited. Nat Rev Nephrol. 2009 May;5(5):270-6. doi: 10.1038/nrneph.2009.43. PMID 19384328
- [Background] Frokiaer J, Marples D, Knepper MA, Nielsen S. Bilateral ureteral obstruction downregulates expression of vasopressin-sensitive AQP-2 water channel in rat kidney. Am J Physiol. 1996 Apr;270(4 Pt 2):F657-68. doi: 10.1152/ajprenal.1996.270.4.F657. PMID 8967344
- [Background] Marples D, Frokiaer J, Dorup J, Knepper MA, Nielsen S. Hypokalemia-induced downregulation of aquaporin-2 water channel expression in rat kidney medulla and cortex. J Clin Invest. 1996 Apr 15;97(8):1960-8. doi: 10.1172/JCI118628. PMID 8621781
- [Background] Bustamante M, Hasler U, Leroy V, de Seigneux S, Dimitrov M, Mordasini D, Rousselot M, Martin PY, Feraille E. Calcium-sensing receptor attenuates AVP-induced aquaporin-2 expression via a calmodulin-dependent mechanism. J Am Soc Nephrol. 2008 Jan;19(1):109-16. doi: 10.1681/ASN.2007010092. Epub 2007 Nov 21. PMID 18032798
- [Background] Procino G, Carmosino M, Tamma G, Gouraud S, Laera A, Riccardi D, Svelto M, Valenti G. Extracellular calcium antagonizes forskolin-induced aquaporin 2 trafficking in collecting duct cells. Kidney Int. 2004 Dec;66(6):2245-55. doi: 10.1111/j.1523-1755.2004.66036.x. PMID 15569313
- [Background] Moeller HB, Rittig S, Fenton RA. Nephrogenic diabetes insipidus: essential insights into the molecular background and potential therapies for treatment. Endocr Rev. 2013 Apr;34(2):278-301. doi: 10.1210/er.2012-1044. Epub 2013 Jan 29. PMID 23360744
- [Background] Patrick L, Uzick M. Cardiovascular disease: C-reactive protein and the inflammatory disease paradigm: HMG-CoA reductase inhibitors, alpha-tocopherol, red yeast rice, and olive oil polyphenols. A review of the literature. Altern Med Rev. 2001 Jun;6(3):248-71. PMID 11410071
- [Result] Bonfrate L, Procino G, Wang DQ, Svelto M, Portincasa P. A novel therapeutic effect of statins on nephrogenic diabetes insipidus. J Cell Mol Med. 2015 Feb;19(2):265-82. doi: 10.1111/jcmm.12422. Epub 2015 Jan 16. PMID 25594563
- [Result] Murer L, Addabbo F, Carmosino M, Procino G, Tamma G, Montini G, Rigamonti W, Zucchetta P, Della Vella M, Venturini A, Zacchello G, Svelto M, Valenti G. Selective decrease in urinary aquaporin 2 and increase in prostaglandin E2 excretion is associated with postobstructive polyuria in human congenital hydronephrosis. J Am Soc Nephrol. 2004 Oct;15(10):2705-12. doi: 10.1097/01.ASN.0000139689.94776.7A. PMID 15466275
- [Result] Procino G, Milano S, Carmosino M, Barbieri C, Nicoletti MC, Li JH, Wess J, Svelto M. Combination of secretin and fluvastatin ameliorates the polyuria associated with X-linked nephrogenic diabetes insipidus in mice. Kidney Int. 2014 Jul;86(1):127-38. doi: 10.1038/ki.2014.10. Epub 2014 Feb 12. PMID 24522493
- [Result] Procino G, Barbieri C, Carmosino M, Rizzo F, Valenti G, Svelto M. Lovastatin-induced cholesterol depletion affects both apical sorting and endocytosis of aquaporin-2 in renal cells. Am J Physiol Renal Physiol. 2010 Feb;298(2):F266-78. doi: 10.1152/ajprenal.00359.2009. Epub 2009 Nov 18. PMID 19923410
- [Result] Procino G. Fluvastatin Increases AQP2 Urine Excretion in a Dyslipidemic Patient with Nephrogenic Diabetes Insipidus: An In Vivo and In Vitro Study. Journal of Diabetes & Metabolism 2014; 5(7); 1000408